CLINICAL TRIAL: NCT01684514
Title: Confocal Laser Endomicroscopy Findings in Patients With Proctosigmoiditis Before and After Initiation of Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, John Gasdal Karstensen, MD, ph.d.-student, Herlev Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H-1-2012-089 sub-1
Record Dates: First submitted 2012-09-06; First posted 2012-09-13 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Colitis, Ulcerative
Keywords: confocal laser endomicroscopy; inflammatory bowel disease; colitis, ulcerative
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- colitis, ulcerative (Experimental): Enrolled patients will be examined by conventional colonoscopy and confocal laser endomicroscopy before and after initiation of topical treatment, respectively.
  Interventions: Device: Confocal laser endomicroscopy
- Control group (Sham Comparator): A control group will be examined by conventional colonoscopy and confocal laser endomicroscopy.
  Interventions: Device: Confocal laser endomicroscopy

INTERVENTIONS:
Device: Confocal laser endomicroscopy — Within recent years a new approach was introduced, wherein the microscopic structures of the intestinal mucous can be evaluated continuously in vivo during the endoscopic procedure. The technique is called confocal laser endomicroscopy (CLE). CLE functions by means of a laser device, which is inserted or build into an endoscope, and used as an illuminator of the lining of a small area and at a precise depth. The tissue is first added with fluorescence by intravenous administration. The reflection of the mucosa is captured in a focused area and magnified by which a two-dimensional image of mucosal microscopic structures is formed. This provides us with an "optical biopsy", which can be compared with a similar microscopic image.

SUMMARY:
Confocal laser endomicroscopy (CLE) is a novel method in evaluation of microscopic structures in vivo. The examination is carried out with a confocal laser endomicroscope, which is either part of the endoscope (manufactured by Pentax) or probe based (manufactured by Cellvizio). Hereby, all parts of the gastrointestinal (GI) tract can be examined. The method has potential to replace conventional microscopy and the dynamic nature of the procedure allows visualization of structures and cellular processes in almost real-time. This provides us with a potentially new diagnostic tool with a promising future. To date only a few studies have been published on inflammatory bowel disease (IBD) and in the literature high-quality research is still lacking.

The project consists of a blinded prospective observation and methodology study including inter- and intra-observation of patients with proctitis before and after initiation of local treatment.

Hypothesis: CLE can be used to assess the degree and extend of acute and chronic inflammation and treatment response in patients with ulcerative colitis and is a sensitive supplementary to conventional diagnostics.

DETAILED DESCRIPTION:
Confocal laser endomicroscopy findings in patients with proctosigmoiditis before and after initiation of treatment

Background Inflammatory bowel disease (IBD) includes Crohn's disease and ulcerative colitis. Crohn's disease often strikes the terminal ileum, but may occur from the mouth to the anus. It is characterized by segmental spreading with transmural inflammation and occasional presence of granulomas in the tissue samples. Ulcerative colitis is only found in the colon and involves in practice always the rectum. The inflammation is limited to the mucosa and submucosa, and the diffusion is continuous.

The development of endoscopy has made these procedures a central part of the diagnostic and therapeutic management of patients with gastrointestinal diseases, including IBD. The entire gastrointestinal tract is now available for inspection and therapy. A limitation of these studies is that the histology, which is often essential for the diagnosis and treatment of the patient, cannot always be precisely evaluated by a conventional examination. The proper handling of detected lesions require in addition to the endoscopic evaluation, a histological evaluation of the tissue involved, making tissue samples necessary in order to obtain a definitive diagnosis and thus optimal handling. Therefore, during the endoscopic procedure tissue samples from the intestinal mucosa must be taken, which rarely involves a greater risk to the patient, but causes a delay, due to preparation time for the histological analysis and in some cases even due to re-examination if histopathology is negative. In the treatment of IBD the endoscopic assessment of the severity and extension is absolutely essential for the choice of treatment. The "Gold standard" for the optimal treatment is called "deep" remission, defined by clinical and endoscopic remission as assessed by conventional endoscopy.

Within recent years a new approach was introduced, wherein the microscopic structures of the intestinal mucous can be evaluated continuously in vivo during the endoscopic procedure. The technique is called confocal laser endomicroscopy (CLE). CLE functions by means of a laser device, which is inserted or build into an endoscope, and used as an illuminator of the lining of a small area and at a precise depth. The tissue is first added with fluorescence by intravenous administration. The reflection of the mucosa is captured in a focused area and magnified by which a two-dimensional image of mucosal microscopic structures is formed. This provides us with an "optical biopsy", which can be compared with a similar microscopic image.

This provides us with a potential opportunity for immediate diagnosing and targeted therapy during the same procedure. The optical biopsy is stored digitally in such a way that it can also be evaluated postprocedure. During CLE multiple frames are generated per second, which is stored continuously, thereby forming a movie sequence, so that the microscopic assessment of the tissue becomes dynamic i.e. the flow in the small vessels may be observed.

A current hypothesis about the pathogenesis of IBD is that a defective barrier function may be a key element. The intestinal barrier is composed of epithelial cells, which are bound together by the so-called "tight junctions". Experimental studies have shown an increased intestinal permeability in IBD patients and that the degree of permeability is a prognostic indicator for the relapse of Crohn's disease. In CLE-studies, the defective barrier function has been identified in vivo as an efflux of fluorescein through the intestinal wall and demonstrated to be significantly greater in IBD patients compared to a healthy control group. The spacing between the epithelial cells are also increased. In patients in remission a defective barrier function predisposes to relapse of their disease. However, it is not possible to realize this dysfunction by a conventional histological examination, as well as other parameters, which require a dynamic microscopic evaluation. By implementing CLE the sensitivity of the endoscopic assessment may increase, which may change not only the characteristics of "deep" remission, but also assessment of the diseases activity.

CLE is at present a rapidly growing field of development which has primarily been used in connection with endoscopy of the digestive tract, but also has been used in connection with endoscopy of the urinary and respiratory tract. CLE have been shown, to reduce the number of tissue samples significantly without compromising the diagnosis. Furthermore, several studies suggest that CLE can contribute to a more accurate diagnosis, and preliminary studies suggest that the degree of the disease can be estimated better compared to conventional endoscopy. Yet, there is no data evaluating the applicability of the method in relation to monitoring of treatment response and as a real prognostic tool. CLE is a new method, and therefore still many unresolved issues and areas to be clarified exist before the technology can finally be implemented in the daily practice.

There is in the research group led by professor of endoscopy Peter Vilmann several years fostered a greater experience in the introduction of new methods. This includes the implementation of relevant studies and the collection and publication of scientific data at an international level, so that the modality can find its proper place for the diagnosis and treatment of patients.

Introduction: By conventional colonoscopy, the degree and spread of inflammation is often underestimated or overlooked in patients with acute inflammation due to insufficient sensitivity. In ulcerative colitis the course of the disease and in particular the risk of treatment failure is related to the degree of acute inflammation, which in addition to clinical and endoscopic observations is assessed by changes in crypt architecture, and infiltration of acute inflammatory cells in the lamina propria. The dissemination of the disease is also particularly important for the choice of treatment, which changes successively from suppositories to enemas and to systemic corticosteroids depending on the proximal boundary of the inflammation. Taking tissue samples may partially prevent underestimation, but this is time consuming, expensive and rarely leads to a radically change of treatment strategy, since endoscopy is the reference in this context. The literature suggest two classifications of inflammation based on CLE, which we partly - and for a start, will use to estimate disease activity before and after initiation of treatment and in a control group. In addition, personal observations will be recorded and analyzed. This assessment will subsequently be used for an intra-and inter-observer study and a stratification of CLE-observations in relation to acute inflammation and degree in tissue samples.

Hypothesis: CLE can be used to assess the degree and extend of acute and chronic inflammation and treatment response in patients with ulcerative colitis and is a sensitive supplementary to conventional diagnostics.

Design: A blinded prospective observation and methodology study in patients before and after initiation of topical steroid treatment with subsequent calculation of intra-and inter-observer variability.

Method: Enrolled patients will be examined by conventional colonoscopy and CLE before and after initiation of topical treatment, respectively. The degree and distribution of acute inflammation will be assessed by conventional microscopy (Mayo score), CLE (crypt architecture, micro vascular changes and the presence of inflammatory cells in the lamina propria and defective barrier function) and histology biopsies. It is expected that not previously described CLE-finding will be found, and that these will be recorded and evaluated as described above.

The terminal ileum and each colonic segment is (caecum, ascending colon, transversal colon, descending colon, colon sigmoid and rectum) assessed as described above. CLE findings will be graded for analysis according to the following scales:

Crypt Architecture: 1: Normal, 2: Changed shape, size and distribution, 3: Crypt destruction and abscess

Micro vascular changes: 1: Normal, 2: Slightly higher in number and moderately dilated, 3: Significantly higher in number and massively dilated

Infiltration of inflammatory cells: 1: No, 2: Presence <50% of the crypts, 3: Presence> 50% of the crypts

Defective barrier function: 1: Normal, 2: Functional defect, 3: Structural defect

The correlation between histology (the "gold standard"), the Mayo score, which is a combined clinical and endoscopic index, and CLE will be calculated. This applies to both IBD patients as the control group. An intra-and inter-observer study is planned after the initial study, where CLE operators are blinded with respect to each other. The pathologist is blinded to conventional and CLE observations. CLE results are stratified in order to identify which of the recorded CLE parameters correlates best with the other two methods, and is therefore most suitable for further studies with focus on inflammation. In addition, a determination of the relationship between CLE findings and the treatment effect for the individual patient is conducted.

Statistical method: Comparison of CLE-findings in relation to the Mayo score and histology is made using Spearman correlation analysis. To evaluate the treatment effect the Wilcoxon Signed Rank test is used. In the inter-and intra-observer study weighted kappa statistics are used.

Patient: A complete sample-size calculation has been made for the inter-and intra-observer study of the individual CLE parameters by 3 observers. If possible, to achieve a kappa value of 0.9 with a confidence interval of 0.05, there must be 122 observations. If we register Mayo score, CLE parameters and take tissue samples for pathology in all the abovementioned intestinal segments during two endoscopies, 14 observations for each patient will be registered which subsequently are assessed in relation to each of the parameters used in the study. If there is no waivers, all ileocolonoscopies are fulfilled and all CLE observations can be analyzed, only 9 patients needs to be included. It is assumed, however, that if only 25% of the expected observations are obtained, since some CLE observations will be unsatisfactory, some examinations will be interrupted, and some patients will only be only evaluated once. Thus, 36 patients must be enrolled in the study to achieve the desired strength, of which 10 are in the control group.

ELIGIBILITY:
Inclusion Criteria:

Patients with active proctitis or proctosigmoiditis due to ulcerative colitis, where an indication for treatment and colonoscopy exists. Newly diagnosed as well as patients already in oral 5-ASA therapy, may be included.

The control group will consist of patients without known or suspected IBD. Patients must be of legal age. Patients who have received written informed consent.

Exclusion Criteria:

Increased p-creatinine and/or demonstrated allergy to fluorescein. Pregnant and lactating women. Ongoing systemic immunosuppressive therapy with prednisolone, azathioprine or biological agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
CLE findings are recorded and compared with the findings of conventional colonoscopy (Mayo score), including observations for the control group | The trial will go on for 2 years
CLE and colonoscopy findings are compared with the pathological evaluation of tissue samples. | The trial will go on for 2 years
Intra-and inter-observer agreement between 3 CLE operators is calculated by kappa statistics | The trial will go on for 2 years

SECONDARY OUTCOMES:
Effect of therapy with topical therapy, based on the results of the conventional colonoscopy and CLE | The trial will go on for 2 years
  A determination of the relationship between CLE findings (the parameters described in the protocol and validated in the inter- and intra-observer study) and conventional colonoscopy findings (Mayo-score) with the treatment effect for the individual patient is conducted. To evaluate the treatment effect the Wilcoxon Signed Rank test is used.
Registering time of the procedure. | The trial will go on for 2 years
Registering possible complications | The trial will go on for 2 years
  Registering possible complications meaning intestinal perforations and bleeding

CONTACTS AND LOCATIONS:
Overall Officials: John G Karstensen, MD, Principal Investigator — Gastroenheden, Herlev Hospital
Locations (2):
- Denmark (2):
  - John Gásdal Karstensen, Birkerød
  - Gastroenheden, Herlev Hospital, Herlev

REFERENCES:
- [Background] Schroeder KW, Tremaine WJ, Ilstrup DM. Coated oral 5-aminosalicylic acid therapy for mildly to moderately active ulcerative colitis. A randomized study. N Engl J Med. 1987 Dec 24;317(26):1625-9. doi: 10.1056/NEJM198712243172603. PMID 3317057
- [Background] Riley SA, Mani V, Goodman MJ, Dutt S, Herd ME. Microscopic activity in ulcerative colitis: what does it mean? Gut. 1991 Feb;32(2):174-8. doi: 10.1136/gut.32.2.174. PMID 1864537
- [Background] Li CQ, Xie XJ, Yu T, Gu XM, Zuo XL, Zhou CJ, Huang WQ, Chen H, Li YQ. Classification of inflammation activity in ulcerative colitis by confocal laser endomicroscopy. Am J Gastroenterol. 2010 Jun;105(6):1391-6. doi: 10.1038/ajg.2009.664. Epub 2009 Nov 24. PMID 19935787
- [Background] Wu K, Liu JJ, Adams W, Sonn GA, Mach KE, Pan Y, Beck AH, Jensen KC, Liao JC. Dynamic real-time microscopy of the urinary tract using confocal laser endomicroscopy. Urology. 2011 Jul;78(1):225-31. doi: 10.1016/j.urology.2011.02.057. Epub 2011 May 23. PMID 21601243
- [Background] Kiesslich R, Goetz M, Neurath MF. Confocal laser endomicroscopy for gastrointestinal diseases. Gastrointest Endosc Clin N Am. 2008 Jul;18(3):451-66, viii. doi: 10.1016/j.giec.2008.03.002. PMID 18674696
- [Background] Fuchs FS, Zirlik S, Hildner K, Frieser M, Ganslmayer M, Schwarz S, Uder M, Neurath MF. Fluorescein-aided confocal laser endomicroscopy of the lung. Respiration. 2011;81(1):32-8. doi: 10.1159/000320365. Epub 2010 Aug 21. PMID 20733287
- [Background] Liu JJ, Wong K, Thiesen AL, Mah SJ, Dieleman LA, Claggett B, Saltzman JR, Fedorak RN. Increased epithelial gaps in the small intestines of patients with inflammatory bowel disease: density matters. Gastrointest Endosc. 2011 Jun;73(6):1174-80. doi: 10.1016/j.gie.2011.01.018. Epub 2011 Mar 11. PMID 21396639
- [Background] Kiesslich R, Duckworth CA, Moussata D, Gloeckner A, Lim LG, Goetz M, Pritchard DM, Galle PR, Neurath MF, Watson AJ. Local barrier dysfunction identified by confocal laser endomicroscopy predicts relapse in inflammatory bowel disease. Gut. 2012 Aug;61(8):1146-53. doi: 10.1136/gutjnl-2011-300695. Epub 2011 Nov 24. PMID 22115910
- [Background] Wyatt J, Vogelsang H, Hubl W, Waldhoer T, Lochs H. Intestinal permeability and the prediction of relapse in Crohn's disease. Lancet. 1993 Jun 5;341(8858):1437-9. doi: 10.1016/0140-6736(93)90882-h. PMID 8099141
- [Background] Peeters M, Ghoos Y, Maes B, Hiele M, Geboes K, Vantrappen G, Rutgeerts P. Increased permeability of macroscopically normal small bowel in Crohn's disease. Dig Dis Sci. 1994 Oct;39(10):2170-6. doi: 10.1007/BF02090367. PMID 7924738
- [Background] Gheorghe C, Cotruta B, Iacob R, Becheanu G, Dumbrava M, Gheorghe L. Endomicroscopy for assessing mucosal healing in patients with ulcerative colitis. J Gastrointestin Liver Dis. 2011 Dec;20(4):423-6. PMID 22187709
- [Background] Wang TD. Confocal microscopy from the bench to the bedside. Gastrointest Endosc. 2005 Nov;62(5):696-7. doi: 10.1016/j.gie.2005.06.002. No abstract available. PMID 16246681
- [Background] Kiesslich R, Goetz M, Lammersdorf K, Schneider C, Burg J, Stolte M, Vieth M, Nafe B, Galle PR, Neurath MF. Chromoscopy-guided endomicroscopy increases the diagnostic yield of intraepithelial neoplasia in ulcerative colitis. Gastroenterology. 2007 Mar;132(3):874-82. doi: 10.1053/j.gastro.2007.01.048. Epub 2007 Jan 31. PMID 17383417
- [Derived] Karstensen JG, Saftoiu A, Brynskov J, Hendel J, Ciocalteu A, Klausen P, Klausen TW, Riis LB, Vilmann P. Confocal laser endomicroscopy in ulcerative colitis: a longitudinal study of endomicroscopic changes and response to medical therapy (with videos). Gastrointest Endosc. 2016 Aug;84(2):279-286.e1. doi: 10.1016/j.gie.2016.01.069. Epub 2016 Mar 2. PMID 26945556